CLINICAL TRIAL: NCT03938467
Title: Effect of Antiseptic Irrigation With 0.05% Chlorhexidine Gluconate (Irrisept) on Incidence of Cutibacterium Acnes in Shoulder Arthroplasty
Brief Title: Irrisept C.Acnes Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Orthopaedic Associates of Michigan, PC (Other)
Collaborators: Mercy Health (Other)
Responsible Party: Principal Investigator, Tim Lenters, Orthopedic Surgeon, Orthopaedic Associates of Michigan, PC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RVO-IRR-2019
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Rate of Positive Culture Growth for C.Acnes From Specimens Obtained From the Shoulders of Patients Undergoing Primary Shoulder Arthroplasty
Keywords: Shoulder Arthroplasty; C.acnes; Cutibacterium acnes; Irrisept

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antiseptic Cleanser (Experimental): Standard prophylaxis will be administered by Irrisept patients as would individuals in the control group. In addition, these Irrisept study subjects will be supplemented with the use of Irrisept irrigation by the study surgeon during the patient's surgical procedure. Standard times for irrigation will include immediately after incision through the dermal layer, and immediately prior to implantation of any prosthetic components. Final irrigation will be performed just prior to closure of the deltopectoral interval.
  Interventions: Drug: Antiseptic Cleanser
- Standard of Care Prophylaxis (No Intervention): Standard prophylaxis includes use of chlorhexidine wipes (Sage cloth) the night before and morning of surgery on the surgical site over the anterior shoulder.

INTERVENTIONS:
Drug: Antiseptic Cleanser — Contains 0.05% Chlorhexidine gluconate in sterile water for irrigation. The mechanical action of the Irrisept system removes bacteria and debris without harming underlying tissues. Irrisept has demonstrated broad spectrum bactericidal activity against antibiotic-resistant strains. Its contents are wrapped in two sequential sterilization wraps which repel water blood, and saline, making it effective against both air and water borne bacteria.
  Other Names: Irrisept Wound Cleansing System
  Arms: Antiseptic Cleanser

SUMMARY:
A Prospective, Randomized, Controlled Trial Comparing An Irrisept Antiseptic Irrigation With 0.05% Chlorhexidine Gluconate versus Standard of Care Prophylaxis Chlorohexidine Wipes

DETAILED DESCRIPTION:
The purpose of this prospective randomized control trial is to access outcomes of positive culture growth of C. acnes from specimens obtained from the shoulders of patients undergoing primary shoulder arthroplasty whose intraoperative management includes Irrisept antiseptic irrigation and compare it to patients whose management includes standard of care prophylaxis wipes.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed the IRB-approved informed consent form specific to this study prior to undergoing any research related procedures
2. Patient can read and understand English
3. Patient who will undergo a primary shoulder arthroplasty
4. Patient is over the age of 18

Exclusion Criteria:

1. Patient who has had a previous surgery on the ipsilateral shoulder
2. Patient has a known allergy to topical iodine or Chlorohexidine gluconate.
3. Patient has had non-surgical prophylaxis antibiotic treatment within 14 days of index surgery
4. Patient requires a revision procedure for a previous ipsilateral shoulder surgery
5. Patient has any significant pathology that, in the opinion of investigator, makes the patient unsuitable for study participation
6. Patient is a pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
C.acnes Growth Rate | 12 months
  To compare the rate of C.acnes using two different antiseptic protocols

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 6 months
  Assessment of clinical/subjective feedback via questionnaires during the postoperative follow up period. VAS assessment: [0 (no pain) - 10 (worse possible pain)]
ROM | 6 Months
  Range of Motion
American Shoulder and Elbow Surgeons Shoulder Score (ASES) | 6 Months
  the Society of the American Shoulder and Elbow Surgeons to facilitate standardization of outcome measures.

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopaedic Associates of Michigan, PC, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horneff JG 3rd, Hsu JE, Voleti PB, O'Donnell J, Huffman GR. Propionibacterium acnes infection in shoulder arthroscopy patients with postoperative pain. J Shoulder Elbow Surg. 2015 Jun;24(6):838-43. doi: 10.1016/j.jse.2015.03.008. PMID 25979553
- [Background] Levy O, Iyer S, Atoun E, Peter N, Hous N, Cash D, Musa F, Narvani AA. Propionibacterium acnes: an underestimated etiology in the pathogenesis of osteoarthritis? J Shoulder Elbow Surg. 2013 Apr;22(4):505-11. doi: 10.1016/j.jse.2012.07.007. Epub 2012 Sep 13. PMID 22981447
- [Background] Matsen FA 3rd, Butler-Wu S, Carofino BC, Jette JL, Bertelsen A, Bumgarner R. Origin of propionibacterium in surgical wounds and evidence-based approach for culturing propionibacterium from surgical sites. J Bone Joint Surg Am. 2013 Dec 4;95(23):e1811-7. doi: 10.2106/JBJS.L.01733. PMID 24306704
- [Background] Matsen FA 3rd, Russ SM, Bertelsen A, Butler-Wu S, Pottinger PS. Propionibacterium can be isolated from deep cultures obtained at primary arthroplasty despite intravenous antimicrobial prophylaxis. J Shoulder Elbow Surg. 2015 Jun;24(6):844-7. doi: 10.1016/j.jse.2014.10.016. Epub 2014 Dec 26. PMID 25547858
- [Background] Mook WR, Klement MR, Green CL, Hazen KC, Garrigues GE. The Incidence of Propionibacterium acnes in Open Shoulder Surgery: A Controlled Diagnostic Study. J Bone Joint Surg Am. 2015 Jun 17;97(12):957-63. doi: 10.2106/JBJS.N.00784. PMID 26085528
- [Background] Sethi PM, Sabetta JR, Stuek SJ, Horine SV, Vadasdi KB, Greene RT, Cunningham JG, Miller SR. Presence of Propionibacterium acnes in primary shoulder arthroscopy: results of aspiration and tissue cultures. J Shoulder Elbow Surg. 2015 May;24(5):796-803. doi: 10.1016/j.jse.2014.09.042. Epub 2014 Dec 4. PMID 25483906
- [Background] Sabetta JR, Rana VP, Vadasdi KB, Greene RT, Cunningham JG, Miller SR, Sethi PM. Efficacy of topical benzoyl peroxide on the reduction of Propionibacterium acnes during shoulder surgery. J Shoulder Elbow Surg. 2015 Jul;24(7):995-1004. doi: 10.1016/j.jse.2015.04.003. PMID 26067191